CLINICAL TRIAL: NCT02175316
Title: Effects of Enhanced External Counterpulsation on Delayed Onset Muscle Soreness, a Pilot Study
Brief Title: Enhanced External Counterpulsation on Delayed Onset Muscle Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FDG20130045H
Record Dates: First submitted 2014-05-21; First posted 2014-06-26 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2017-09

CONDITIONS: Muscle Tightness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental: EECP for DOMS (Experimental): All enrolled subjects will receive EECP treatment Delayed Onset Muscle Soreness.
  Interventions: Device: Enhanced External Counterpulsation

INTERVENTIONS:
Device: Enhanced External Counterpulsation — Enhanced External Counterpulsation
  Other Names: Lumenair Enhanced External Counterpulsation Therapy System, Vasomedical

SUMMARY:
This study will evaluate the effects of Enhanced External Counterpulsation on delayed onset muscle soreness. The primary outcomes will be duration of delayed onset muscle soreness, WBC count, CRP count, CPK count, and pain tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy active Duty or DoD beneficiaries between 25 and 59 years old

Exclusion Criteria:

* Not on a physical profile
* Not taking any OTC or prescription pain medications or workout supplements

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07-25 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Change in delayed onset muscle soreness over time. | At 3, 6, 9, 12, 15, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48 Hours
  Likert pain surveys

SECONDARY OUTCOMES:
Pain tolerance | Baseline, 24 hours, 2 days 3 days 4 days 33 days
  Pain tolerance measured by mmHg pressure required to elicit a delayed-onset muscle pain response.
Bio-markers for muscle inflammation | Baseline, 24 hours, 2 days 3 days 4 days 33 days
  Bio-markers for muscle inflammation: C-reactive protein, creatine phosphokinase, and white blood cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Shah, Principal Investigator — United States Air Force
Locations (1):
- David Grant USAF Medical Center, Travis Air Force Base, California, United States